CLINICAL TRIAL: NCT02572154
Title: Male Factor in Early Recurrent Pregnancy Loss : Study of Sperm DNA Fragmentation in Patients With Unexplained Recurrent Pregnancy Loss.
Brief Title: Sperm DNA Fragmentation in Recurrent Pregnancy Loss
Acronym: PARTHOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11 198 08
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2016-10

CONDITIONS: RECURRENT PREGNANCY LOSS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cases (Other): men from couples with RPL after natural pregnancies, had blood and sperm samples for sperm DNA fragmentation exploration
  Interventions: Other: Blood and sperm samples
- Controls (Other): men from couples who have a child consequently to a natural pregnancy, had blood and sperm samples for sperm DNA fragmentation exploration
  Interventions: Other: Blood and sperm samples

INTERVENTIONS:
Other: Blood and sperm samples — 20 ml of blood and sperm samples for sperm DNA fragmentation exploration

SUMMARY:
In human, 2% of couples experimented Recurrent pregnancy loss (RPL). Currently, while etiological investigations were performed, 40 to 50 % of RPL were unexplained. In animals' studies, several studies have underlined the importance of sperm quality for a normal embryo development. In human, epidemiological studies have demonstrated that several male risk factors have effects on development (male mediated development toxicology). However, few studies have explored sperm DNA fragmentation on embryo development but after in vitro fertilization. In natural pregnancy only rare studies have been performed but with different populations definitions and different methods of sperm exploration. In this context sperm DNA fragmentation exploration appears justified. The present study purpose to conduct a case - control study in order to research paternal role in RPL.

ELIGIBILITY:
Inclusion Criteria:

* Cases: Man from couples with RPL (more than 2 miscarriages) RPL classical etiological exploration negative (unexplained RPL) Healthy voluntaries
* Control: Man from couples who have a child after a natural pregnancy obtained in the year following child desire.

Healthy voluntaries

Exclusion Criteria:

* Cases: Etiological exploration of RPL positive Man with chromosomal anomaly
* Cases and controls:

Ongoing pathology Chemotherapy or radiotherapy history Hyperthermia (fever) in the last three months Pregnancy obtained by assisted reproduction (Inseminations, in vitro fertilization) Women > 38 year old

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
sperm DNA fragmentation | baseline
  Percentage of sperm with fragmented DNA in both groups

SECONDARY OUTCOMES:
Sperm aneuploidy | baseline
  Percentage of spermatozoa with aneuploidy.
Sperm Volume | baseline
Sperm pH | baseline
sperm concentration | baseline
sperm concentration of round cells | baseline
percentage of motile and morphologically normal spermatozoa in sperm | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bujan, PUPH, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - Chu Bordeaux, Bordeaux
  - APHM, Marseille
  - Chu Toulouse, Toulouse

REFERENCES:
- [Result] Esquerre-Lamare C, Walschaerts M, Chansel Debordeaux L, Moreau J, Bretelle F, Isus F, Karsenty G, Monteil L, Perrin J, Papaxanthos-Roche A, Bujan L. Sperm aneuploidy and DNA fragmentation in unexplained recurrent pregnancy loss: a multicenter case-control study. Basic Clin Androl. 2018 Apr 2;28:4. doi: 10.1186/s12610-018-0070-6. eCollection 2018. PMID 29619224